CLINICAL TRIAL: NCT03227315
Title: Is There a Relationship Between Stress Tolerance and Analgesic Consumption in Obese Patients?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hakan Tapar, Assist.Prof, Tokat Gaziosmanpasa University
Other Study IDs: 17-KAEK-077
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Distress Tolerance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preoperative anxiety level of patients affects postoperative analgesic consumption. However, there were no studies that showed a relationship between the level of stress tolerance and analgesic consumption in the literature. In this study, investigators wanted to investigate the effect of stress tolerance on analgesic consumption of patient.

DETAILED DESCRIPTION:
After approval, patients enrolled in the study is invited to complete the Pain Catastrophizing Scale questionnaire, Distress Tolerance Scale and Beck anxiety scale.After surgery, VAS scores of the patients will be evaluated (in the recovery room, 2,6,12 and 24 hours). and patients with VAS> 3 will receive 2 mg of morphine.The relationship between total analgesic consumption and the stress tolerance will be evaluated.The study will be performed with 69 sleeve gastrectomy patients(BMI>30).

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 60 years
* Planned to sleeve gastrectomy
* An American Society of Anesthesiologists score of 1 or 2 BMI>30

Exclusion Criteria:

* Psychiatric diseases
* Rejected to participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The Patients that will happen sleeve gastrectomy
Sampling Method: Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2017-11-20 (Estimated); Study Completion 2017-12-10 (Estimated)

PRIMARY OUTCOMES:
The effect of patient anxiety tolerance on analgesic consumption | one time in four months
  Assessment of analgesic consumption according to the patient's anxiety. tolerance.The distress tolerance scale will be used for this.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Tapar, Principal Investigator — Gaziosmanpasa university
Locations (2):
- Turkey (Türkiye) (2):
  - Gaziosmanpasa University, Tokat Province
  - Hakan Tapar, Tokat Province

IPD SHARING:
Plan to Share IPD: No